CLINICAL TRIAL: NCT04167995
Title: Assessment of Probiotic Strain Lactobacillus Acidophilus LB Supplementation as Adjunctive Management of Attention-deficit Hyperactivity Disorder in Children and Adolescents: a Randomized Controlled Clinical Trial
Brief Title: Assessment of Probiotics Lactobacillus in the Management of Attention Deficit Hyperactive Disorder
Acronym: ADHD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Reham Ibrahim, Associate professor of pediatrics Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWA 000017
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Inattentive; Hyperactivity; Impulsivity
Keywords: Hyperactivity; Inattention; Probiotics
MeSH Terms: conditions — Spasm; Impulsive Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Using a computer-based randomization program. The allocation was concealed in sealed envelopes. Only the researchers collecting and analyzing the data were blinded to the study groups (assessor-blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with attention deficit hyperactive disorser (Active Comparator): patients (n=40) will receive probiotic preparation twice daily (Lacteol Forte; Rameda, Egypt) as sachets containing 10 billion colony forming units (CFU) of Lactobacillus fermentum and Lactobacillus delbruekii for 12 weeks added to standard treatment
  Interventions: Drug: Probiotic Formula lacteal forte
- ADHD not receiving probiotics (No Intervention): ADHD patient (40) on standard treatment

INTERVENTIONS:
Drug: Probiotic Formula lacteal forte — Active Comparator: Patient with attention deficit hyperactive disorder patients (n=40) will receive probiotic preparation twice daily (Lacteol Forte; Rameda, Egypt) as sachets containing 10 billion colony forming units (CFU) of Lactobacillus fermentum and Lactobacillus delbruekii for 12 weeks .
  Other Names: Lacteal forte
  Arms: Patient with attention deficit hyperactive disorser

SUMMARY:
ADHD is a neurodevelopmental disorder characterized by persistent symptoms of inattention and/or hyperactivity and impulsivity that are present before age 18. These symptoms must be evident across ADHD treatment is currently based on a multimodal approach with the combination of psychotherapy and pharmacotherapy, but no reliable markers of treatment response have been identified yet and 20-35% of subjects in clinical trials may have an inadequate response to the treatment The gut microbiome refers to the microbial ecosystem found in the gastrointestinal system of the human species Probiotics are a type of beneficial bacteria that improve health and facilitate intestinal microbial balance Increasing evidence suggests that the gut microbiota plays a key role in the gut-brain communication axis by influencing metabolism, inflammation, the hypothalamic-pituitary-adrenal axis, and neurotransmission multiple domains and cause Impairment in functioning in order to meet the diagnostic criteria for ADHD

DETAILED DESCRIPTION:
All patients will be randomly distributed into two equal groups using a random number generator from computer-based randomization software. the probiotic group (n=40) received probiotic preparation twice daily (Lacteol Forte; Rameda, Egypt) as sachets containing 10 billion colony-forming units (CFU) of Lactobacillus fermentum and Lactobacillus delbruekii for 12 weeks added to a weight-dependent dose of standard treatment (Atomoxetine), and the 40 patients in the control group will not receive the probiotic and on a weight-dependent dose of atomoxetine.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 16 years old.
* Children fulfilled DSM(V) Criteria for ADHD syndrome.

Exclusion Criteria:

* Intelligence quotient (IQ) less than 80% .
* Presence of other medical conditions as chronic medical or neuropsychiatric disorders e.g diabetes mellitus, epilepsy…..etc. hearing or visual impairment, or medications side effects.
* currently taking probiotics or antibiotics

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Conner's Parent Rating Scales-Revised (CRS-R):for follow up | 3 months
  This tool is used in order to assess the profile and severity of symptoms, response to treatment and follow up studies. Items are scored on 14 subscales of symptoms including opposition, cognitive problems, inattention, and hyperactivity.It is usually considered normal when T-scores are less than 60, while scores above 60 are signs of academic, behavioral, or social issues. There are several different classes as well
Child behavior checklist | 3 months
  Parent form to asses the associated internalizing and externalizing behaviour

SECONDARY OUTCOMES:
Conners Continuous Performance Test (CPT) | 3 months
  To asses sustained attention and impulsivity
Wisconsin (Berg) Card Sort Test (WCST) | 3 months
  To evaluate executive function

CONTACTS AND LOCATIONS:
Overall Officials: Reham Ibrahim, Study Director — Ain Shams University
Locations (1):
- Reham Ibrahim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elhossiny RM, Elshahawy HH, Mohamed HM, Abdelmageed RI. Assessment of probiotic strain Lactobacillus acidophilus LB supplementation as adjunctive management of attention-deficit hyperactivity disorder in children and adolescents: a randomized controlled clinical trial. BMC Psychiatry. 2023 Nov 9;23(1):823. doi: 10.1186/s12888-023-05324-4. PMID 37946220